CLINICAL TRIAL: NCT06958081
Title: Acute Effects of Transcranial Direct Current Stimulation on Technical, Expressive, and Scenic Aspects of Musical Performance in Young Orchestra Instrumentalists: A Proof-of-Concept Study
Brief Title: tDCS and Musical Performance in Young Orchestra Musicians
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Principal Investigator, Frederico Barreto Kochem, Principal Investigator and Professor at Centro Universitário Augusto Motta (UNISUAM), Centro Universitário Augusto Motta
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 88146925.0.0000.5235
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Musical Performance; Neuromodulation; Performance Anxiety
Keywords: tDCS; Transcranial Direct Current Stimulation; Music Performance; Motor Control; Self-Efficacy; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an active tDCS group or a sham stimulation group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcome assessors will be blinded to group assignment until the end of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive active transcranial direct current stimulation (tDCS) with a 2.0 mA anodal current applied over the supplementary motor area (FCz) and cathodal electrode over Fp2 for 30 minutes.
  Interventions: Device: Active transcranial direct current stimulation (tDCS)
- Sham tDCS (Sham Comparator): Participants will receive sham transcranial direct current stimulation (tDCS) with the same electrode placement as the active group; however, the current will be turned off after 30 seconds to simulate the initial sensations without delivering prolonged stimulation.
  Interventions: Device: Sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Active transcranial direct current stimulation (tDCS) — 2.0 mA anodal stimulation applied over FCz with cathode over Fp2 for 30 minutes using a transcranial direct current stimulation device.
  Arms: Active tDCS
Device: Sham transcranial direct current stimulation (tDCS) — Sham stimulation mimicking the sensations of tDCS; the current will be turned off after 30 seconds while maintaining electrode placement over FCz and Fp2.
  Arms: Sham tDCS

SUMMARY:
The goal of this clinical trial is to learn if transcranial direct current stimulation (tDCS) can improve the technical, expressive, and stage aspects of musical performance in young orchestra musicians aged 18 to 30 years. The main questions it aims to answer are:

* Does active tDCS improve musical performance compared to sham stimulation?
* Does active tDCS reduce music performance anxiety and increase musical self-efficacy? Researchers will compare the active tDCS group to the sham stimulation group to see if active stimulation has positive effects on musical performance and psychological factors.

Participants will:

* Receive either active or sham tDCS stimulation
* Perform a musical piece before and after stimulation
* Complete questionnaires about anxiety and musical self-confidence

DETAILED DESCRIPTION:
This randomized pilot study aims to investigate the acute effects of transcranial direct current stimulation (tDCS) on the technical, expressive, and stage aspects of musical performance in young orchestra instrumentalists.

A total of 24 musicians, aged 18 to 30 years, with at least three years of orchestral experience, will be randomly assigned to either an active tDCS group or a sham stimulation group. The stimulation will target the supplementary motor area (SMA) using a 2.0 mA anodal current for 30 minutes, with the cathode placed over Fp2. The sham group will undergo the same electrode placement, but the current will be turned off after 30 seconds.

The study will adopt a double-blind design, where neither participants, care providers, investigators, nor outcome assessors will know the group allocations. Each participant will perform a standardized musical piece before and after the intervention, and after a 2-hour interval post-intervention. Performances will be recorded and evaluated by independent expert judges using the Rubric for the Assessment of Music Performance Achievement.

Psychometric evaluations will be conducted using the Mazzarolo Music Performance Anxiety Scale (M-MPAS) and the General Musical Self-Efficacy Scale. Self-assessments of performance and sensations during stimulation will also be collected. Data analysis will compare changes in musical performance, anxiety, and self-efficacy between groups.

This study seeks to provide preliminary evidence on the potential of tDCS to enhance musical performance and psychological factors such as performance anxiety and self-confidence among young musicians. Safety and feasibility of the intervention will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Musicians aged 18 to 30 years.
* Minimum of 3 years of orchestral performance experience.
* Active participation in a stable orchestra or ensemble.
* No history of neurological or psychiatric disorders.
* Not currently using psychotropic medications or recreational drugs.
* Willingness to participate in all study sessions.
* Signed informed consent form.

Exclusion Criteria:

* Presence of metallic implants in the head (e.g., cranial pins, aneurysm clips).
* Presence of implanted electronic devices (e.g., pacemaker).
* History of epilepsy or seizures.
* Prior experience with transcranial direct current stimulation (tDCS).
* Scalp dermatitis or lesions at the electrode placement sites.
* Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Musical Performance Scores (Rubric for the Assessment of Music Performance Achievement) | Baseline, immediately after intervention, and 2 hours after intervention
  Musical performance will be evaluated by independent expert judges using a standardized rubric assessing technical, expressive, and stage presence aspects.

SECONDARY OUTCOMES:
Change in Self-Reported Musical Performance Score (0-10 scale) | Baseline, immediately after intervention, and 2 hours after intervention
  Participants will self-rate the quality of their musical performance on a 0 (worst) to 10 (best) scale after each recording session.
Music Performance Anxiety (Mazzarolo Music Performance Anxiety Scale - M-MPAS) | Baseline
  Participants' levels of music performance anxiety will be assessed using the Mazzarolo Music Performance Anxiety Scale (M-MPAS), a validated 5-item instrument designed to measure cognitive, somatic, and behavioral symptoms of performance anxiety in musicians. Each item is rated on a 7-point Likert scale (0-6), with a total score range from 0 to 30 points. Higher scores indicate greater levels of anxiety, with scores ≥11 suggesting a tendency toward elevated performance anxiety.
Musical Self-Efficacy (General Musical Self-Efficacy Scale) | Baseline
  Musical self-efficacy will be assessed using the performance subscale of the General Musical Self-Efficacy Scale, composed of 11 items rated on a 7-point Likert scale ranging from 1 ("Strongly disagree") to 7 ("Strongly agree"). The total score ranges from 11 to 77, with higher scores indicating greater self-efficacy in musical performance contexts.
Perception of Intervention Received (Active or Sham) | Immediately after intervention
  Participants will report whether they believe they received active stimulation or sham stimulation, to assess effectiveness of blinding.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Galhardoni, Ph.D, Principal Investigator — Neuromodulação em Foco; Renato Santos de Almeida, Ph.D, Study Chair — Centro Universitário Augusto Motta; Débora Cristina Lima da Silva, Ph.D, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro Universitário Augusto Motta (UNISUAM), Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It has not yet been determined whether individual participant data (IPD) will be shared. The decision will depend on future analyses, data sensitivity considerations, and publication plans.

REFERENCES:
- [Background] Álvarez-Díaz M, Muñiz-Bascón LM, Soria-Alemany A, Veintimilla-Bonet A, Fernández-Alonso R. On the design and validation of a rubric for the evaluation of performance in a musical contest. International Journal of Music Education. 2021;39(1):66-79. doi:10.1177/0255761420936443
- [Background] Mazzarolo I, Schubert E. A Short Performance Anxiety Scale for Musicians. Front Psychol. 2022 Jan 26;12:781262. doi: 10.3389/fpsyg.2021.781262. eCollection 2021. PMID 35153903
- [Background] Sanchez-Kuhn A, Perez-Fernandez C, Canovas R, Flores P, Sanchez-Santed F. Transcranial direct current stimulation as a motor neurorehabilitation tool: an empirical review. Biomed Eng Online. 2017 Aug 18;16(Suppl 1):76. doi: 10.1186/s12938-017-0361-8. PMID 28830433
- [Background] Anic A, Olsen KN, Thompson WF. Investigating the Role of the Primary Motor Cortex in Musical Creativity: A Transcranial Direct Current Stimulation Study. Front Psychol. 2018 Oct 1;9:1758. doi: 10.3389/fpsyg.2018.01758. eCollection 2018. PMID 30327622
- [Background] Chinzara TT, Buckingham G, Harris DJ. Transcranial direct current stimulation and sporting performance: A systematic review and meta-analysis of transcranial direct current stimulation effects on physical endurance, muscular strength and visuomotor skills. Eur J Neurosci. 2022 Jan;55(2):468-486. doi: 10.1111/ejn.15540. Epub 2022 Jan 6. PMID 34904303
- [Background] Bikson M, Grossman P, Thomas C, Zannou AL, Jiang J, Adnan T, Mourdoukoutas AP, Kronberg G, Truong D, Boggio P, Brunoni AR, Charvet L, Fregni F, Fritsch B, Gillick B, Hamilton RH, Hampstead BM, Jankord R, Kirton A, Knotkova H, Liebetanz D, Liu A, Loo C, Nitsche MA, Reis J, Richardson JD, Rotenberg A, Turkeltaub PE, Woods AJ. Safety of Transcranial Direct Current Stimulation: Evidence Based Update 2016. Brain Stimul. 2016 Sep-Oct;9(5):641-661. doi: 10.1016/j.brs.2016.06.004. Epub 2016 Jun 15. PMID 27372845